CLINICAL TRIAL: NCT00373243
Title: An Open-label, Non-randomised Study of 20 mg GW406381 Single Dose Pharmacokinetics in Healthy Subjects and in Volunteers With Moderate Hepatic Impairment
Brief Title: A Study Of GW406381 In Volunteers With Moderate Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CXA100754
Record Dates: First submitted 2006-09-05; First posted 2006-09-07 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Pain
Keywords: hepatic impairment pharmacokinetics
MeSH Terms: conditions — Pain | interventions — GW406381X

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subjects receiving GW406381 (Experimental): Subjects will receive single oral dose of 20 milligram (mg) of GW406381.
  Interventions: Drug: GW406381

INTERVENTIONS:
Drug: GW406381 — GW406381 will be available as 10 mg hard gelatin capsules. Subjects will receive two capsules of 10 mg to make 20 mg dose.

SUMMARY:
This study will assess the pharmacokinetics and tolerability of a single dose of GW406381 in subjects with moderate hepatic impairment in comparison to matched healthy volunteers. The hepatically impaired and healthy groups will be given a single 20 mg oral dose of GW406381. Blood samples for PK analysis will be collected pre-dose and over the 72 hours post dosing. Subjects will be housed from the evening before dosing until 24 hours after dosing. A follow-up visit will be conducted between 7 to 10 days from the last dose of study drug.

ELIGIBILITY:
Inclusion criteria:

* Healthy subjects or subjects with moderate hepatic impairment as defined by a Child-Pugh score of 7-9
* Body weight less = 100 kg
* Body mass index (BMI) within range of 19 - 32 32kg/m2

Exclusion criteria:

* Presence of any other significant disease
* Use of any medication within the 2 weeks prior to dosing, unless approved by both the investigator and GSK personnel

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-10-19 (Actual); Primary Completion 2006-09-26 (Actual); Study Completion 2006-09-26 (Actual)

PRIMARY OUTCOMES:
GW406381 pharmacokinetic parameters AUC and Cmax | throughout the study

SECONDARY OUTCOMES:
GW406381 pharmacokinetic parameters Tmax, Total plasma clearance, and if data permits the t1/2 of GW406381 GW404347 pharmacokinetic parameters AUC and Cmax Ex vivo protein binding Clinical laboratory values, adverse events, vital signs and 12 lead ECG | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Hungary (2):
  - GSK Investigational Site, Balantonfured
  - GSK Investigational Site, Budapest

REFERENCES:
- See also: Results for study CXA100754 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/CXA100754?search=study&search_terms=CXA100754#rs